CLINICAL TRIAL: NCT04153097
Title: Real World Observational Study of Pembrolizumab for Chinese Advanced NSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: ZYHX-001
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- pembrolizumab-treated advanced NSCLC: Patients with advanced non-small cell lung cancer treated with pembrolizumab

SUMMARY:
This observational study is designed to assess the efficacy and safety of pembrolizumab for the treatment of Chinese advanced NSCLC.

DETAILED DESCRIPTION:
Pembrolizumab is a humanized antibody used in cancer immunotherapy.The NMPA(China) approved pembrolizumab for first-line treatment of certain patients with advanced NSCLC.

This is a multi-center non-interventional study, advanced NSCLC patients who treated with pembrolizumab and provide written informed consent will be included. The main objective of this study is to evaluate pembrolizumab efficacy and safety in the clinical practice and explore the prognosis-relevant factors of advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of advanced or metastatic NSCLC
2. Patients who receive pembrolizumab for advanced NSCLC.
3. Patients who provided written informed consent.

Exclusion Criteria:

1.Patients who would join any interventional clinical studies from first diagnosis to the end of the pembrolizumab treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total 500 patients who receive pembrolizumab for advanced NSCLC will be enrolled. The patients should be registered consecutively in each site.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-07-30 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Median Overall survival (OS) since start of pembrolizumab | 3 years
  OS was defined as the length of time from the administration of the first-dose until death from any cause.
Objective Response Rate (ORR) since start of pembrolizumab | 6 months
  ORR was defined as the percentage of patients with complete response (CR) and partial response (PR) according to irRECIST.
Rate of Adverse Drug Reaction (ADR) since start of pembrolizumab | up to 3 months after the last dose
  Drug related AEs were evaluated using NCI-CTCAE v5.0

SECONDARY OUTCOMES:
Median Progression Free Survival (PFS) since start of pembrolizumab | 12 months
  PFS is defined as the time from the start of first-dose to first progression disease (PD) or death, whichever is earlier.
Median Time To Treatment failure (TTF) since start of pembrolizumab | 12 months
  TTF is defined as the time from the start of first-dose to discontinuation for any reason, including disease progression, treatment toxicity, patient preference, or death.

CONTACTS AND LOCATIONS:
Overall Officials: Jianying Jianying, MD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (8):
- China (8):
  - The First Affiliated Hospital of College of Medicine Zhejiang University, Hangzhou, Zhejiang
  - Second Affiliated Hospital, Zhejiang University of Medicine, Hangzhou, Zhejiang
  - the First Hospital of Jiaxing, Jiaxing, Zhejiang
  - Jinhua Guangfu Hospital, Jinhua, Zhejiang
  - Ningbo Medical Center Lihuili Eastern Hospital, Ningbo, Zhejiang
  - Quzhou People's Hospital, Quzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The People's Hospital of Zhuji, Zhuji, Zhejiang

IPD SHARING:
Plan to Share IPD: No
No plan to share date of the trial